CLINICAL TRIAL: NCT07116044
Title: Assessment of Response and Impact on Safety, Adherece Anc Persistent During Treatment in an Observational Trial for the Evaluation of the Long-term Effectiveness of Bulevirtide in Patients With Chronic Delta Hepatitis: the ARISTOTELE Study
Brief Title: Assessment of Response and Safety of Bulevirtide Treatment in Patients With Chronic Delta Virus Infection
Acronym: ARISTOTLE
Status: Completed | Type: Observational
Sponsor: University of Molise (Other)
Responsible Party: Principal Investigator, Luca Rinaldi, Associate Professor, University of Molise
Other Study IDs: ARISTOTLE Research Project; Gilead Sciences srl (Other: Università degli Studi del Molise)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Evaluate Response to Treatment Both Biochemically and Virologically to Determine the Safety and Effectiveness of Bulevirtide Therapy in HDV Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: virological tests diagnostic tests — The parameters collected will include blood sugar, HbA1c, complete blood count, lipid profile (total cholesterol, LDL, HDL, triglycerides), liver profile (ALT, AST, total and fractionated bilirubin, alkaline phosphatase, GGT) and renal profile (creatinine, azotemia), electrophoretic protein picture. Additionally, specific data for HDV and HBV infection will be collected, including HBsAg, anti-HBs, anti-HBc, HBV-DNA, and HDV-RNA. The glomerular filtration rate shall be calculated using the formula CKD-EPI.
  • Instrumental Tests: Results of abdominal ultrasounds, Fibroscan®/CAP for the evaluation of liver fibrosis

SUMMARY:
1. The study is non-interventional, multicenter, non-profit
2. The primary objective of the study is to evaluate the safety and efficacy in clinical practice of the drug Bulevirtide in the treatment of patients with chronic HDV hepatitis. The drug is already approved and indicated in the treatment of patients with the aforementioned infectious pathology.
3. The Coordinating Center and the Principal Investigator of the study in question will be, respectively, the Department of Medical Health Sciences "V. Tiberio" and the undersigned Prof. Luca Rinaldi in cooperation with the Azienda dei Colli, Cotugno Hospital in Naples, Dr Antonio Izzi.
4. As regards the further economic aspects, it is underlined that no compensation of any kind is foreseen for the subjects participating in the study and that there are no expenses borne by the subjects participating in the study. The study will be coordinated, managed and analyzed independently.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HDV and HBV-related liver disease considered suitable for antiviral or immunomodulatory treatment.

  * Absence of contraindications to the use of Bulevirtide
  * Age over 18 years.
  * Patients born to therapy or already undergoing cycles of therapy with standard interferon or pegylated.
  * Informed consent to study participation

Exclusion Criteria:

* Specific contraindications to bulevirtide • Presence of decompensated liver disease or other conditions that may interfere with study participation or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HDV and HBV-related liver disease considered suitable for antiviral or immunomodulatory treatment
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of bulevirtide | 12 months
  Evaluate the virological response to treatment with bulevirtide, measured as reduction or clearance of serum or plasma HDV-RNA, after 12 months of treatment.

SECONDARY OUTCOMES:
Maintenance and Adherence to Therapy | 12 months
  Monitor patients' adherence to the bulevirtide treatment regimen, evaluating continuity of treatment and compliance with the prescribed dosage. This includes analysis of any interruptions or changes to treatment and the underlying reasons

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli studi del molise, Campobasso, Seleziona, Italy

IPD SHARING:
Plan to Share IPD: No
e-identified individual ATIs (raw or derived) of study participants
  Additional documentation (protocol, statistical analysis plan, data dictionary